CLINICAL TRIAL: NCT00154778
Title: An Open,Multi-Center,Phase II Clinical Trial tO Evaluate Efficacy and Safety oF TAXOL(PACLITAXEL),UFT,and LEUCOVORIN in Patients With Advanced Gastric Cancer
Brief Title: Taxol(Paclitaxel),UFT and Leucovorin in Patients With Advanced Gastric Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Taipei Veterans General Hospital, Taiwan (Other Government); Tri-Service General Hospital (Other); Mackay Memorial Hospital (Other); National Cheng-Kung University Hospital (Other); National Health Research Institutes, Taiwan (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 910703
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2007-07-31 (Estimated); Status verified 2005-07

CONDITIONS: Gastric Cancer
Keywords: Combination,Chemotherapy,Advanced Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Experimental)
  Interventions: Drug: Taxol, UFT,Leucovorin

INTERVENTIONS:
Drug: Taxol, UFT,Leucovorin

SUMMARY:
The purpose of this study is to evaluate the response rate of Paclitaxel combination chemotherapy with UFT and Leucovorin in patients with advanced gastric cancer.

DETAILED DESCRIPTION:
Since 1982,cancer has been the leading cause of death in Taiwan. In particular,gastric cancer is the fourth leading cause of death in male cancer patients and the sixth for female patients in 2000,accounting for an estimated 2,374 deaths. In recent years, the treatment of gastric cancer patients has gradually been improving due to advances in early diagnosis and surgical techniques. Although chemotherapy and radiation therapy have been used in either the adjuvant or palliative setting, their values are still limited due to their unacceptable toxicity or inadequate efficiency.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years old
2. Patients with histologically confirmed gastric adenocarcinoma, defined as locally advanced unresectable or metastatic or recurrent disease
3. Patients with at least one measurable lesion
4. ECOG performance status of 0,1 or 2
5. Patients with no prior chemotherapy and radiotherapy for metastatic disease (patients who have received and completed prior adjuvant chemotherapy at least 6 months prior to study enrollment may be enrolled into the study, prior taxane chemotherapy should be excluded)
6. Patients with physiological functions (bone marrow, heart, liver, kidney, etc.) meeting the following criteria: WBC >4000/mm3, ANC >1500/mm3, PLT >100,000/mm3, Hb >9.0g/dL, ALT<3 times the ULN (<5 times the ULN for liver metastasis cases), Total bilirubin <1.5mg/dL, Creatinine <the upper limit of normal
7. Accessible for treatment and follow-up
8. Give written informed consent
9. Women of child bearing potential must have a negative plasma or urine pregnancy test within 72 hours prior to start of the study medication

Exclusion Criteria:

1. Patients who received surgery within 14 days prior to enrollment
2. Patients with CNS metastasis
3. History of hypersensitivity related to the administration of polyoxyethylated-castor-oil (cremophor EL)-containing preparation (e.g. cyclosporin,etc.) or hardened-castor-oil-containing preparation (e.g. vitamin preparation for injection,etc.)
4. Patients with a history of severe hypersensitivity
5. Active infectious symptoms
6. Patients with active gastrointestinal bleeding, intestinal obstruction or other situation that dose not allow oral intake of medication
7. Patients with ascites that adversely affects performance status
8. Pre-existing CTC Grade 2 or greater neuropathy (motor or sensory)
9. Pregnant or nursing females
10. Patients who have participated in other clinical trials within 30 days prior to the first dose of the study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2003-03; Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
To evaluate the response rate | 2003~2004

SECONDARY OUTCOMES:
To determine time to progression and safety | 2004~2005

CONTACTS AND LOCATIONS:
Overall Officials: Kun-Huei Yeh, M.D.,Ph.D., Principal Investigator — Department of Oncology, National Taiwan University Hospital
Locations (1):
- Department of Oncology, Nationa Taiwan University Hospital, Taipei, Taipei, Taiwan

REFERENCES:
- [Result] Chao Y, Li CP, Chao TY, Su WC, Hsieh RK, Wu MF, Yeh KH, Kao WY, Chen LT, Cheng AL. An open, multi-centre, phase II clinical trial to evaluate the efficacy and safety of paclitaxel, UFT, and leucovorin in patients with advanced gastric cancer. Br J Cancer. 2006 Jul 17;95(2):159-63. doi: 10.1038/sj.bjc.6603225. Epub 2006 Jun 27. PMID 16804524
- See also: An open, multi-centre, phase II clinical trial to evaluate the efficacy and safety of paclitaxel, UFT, and leucovorin in patients with advanced gastric cancer. — http://www.ncbi.nlm.nih.gov/sites/entrez?cmd=Search&db=PubMed&term=16804524